CLINICAL TRIAL: NCT06054308
Title: Mesothelin-targeted CAR-T Cells as a Neo-adjuvant Treatment in Patients With Resectable Pancreatic Cancers: a Feasibility Study
Acronym: CART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain Clinical Trial Certificate due to tech Unable to obtain Clinical Trial Certificate due to technical difficulties
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The Chinese University of Hong
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSLN CART (Experimental): Endoscopic ultrasound guided injection of mesothelin-targeted CAR-T cells
  Interventions: Other: MSLN CART

INTERVENTIONS:
Other: MSLN CART — Endoscopic ultrasound guided injection of mesothelin-targeted CAR-T cells

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is a cancer of grave prognosis, with only about 10% of patients alive at 5 years after diagnosis. Primary surgical resection is feasible in about 10-15% of patients with an early-stage disease. Another 30-35% of patients have locally advanced disease with invasion into major vasculature but without detectable metastases. Surgery offers a chance of cure. The introduction of adjuvant multi-agent chemotherapy has improved prognosis after surgery.

In the management of patients with PDAC, the role of neoadjuvant therapy is less certain. Neoadjuvant therapy for pancreatic cancer can in theory control early systemic spread and improve rate of having no macroscopic or microscopic residual tumor (R0 resection). In the The European Study Group for Pancreatic Cancer (ESPAC-5) study, neoadjuvant combination chemotherapy did not increase rate of resection who had borderline-resectable disease but appears to improve overall survival (OS).

Chimeric antigen receptor (CAR) T-cell therapy may represent a new paradigm in the treatment of pancreatic cancer. Mesothelin (MSLN) is a 40 kDa membrane protein not expressed in normal cells, but highly expressed in a variety of cancer cells, such as mesothelioma, lung, breast, ovarian, gastric and pancreatic cancer. MSLN is expressed about 80% of PDAC.

There are several immunotherapies targeting MSLN for PDAC treatment, including antibody-based drugs (monoclonal antibodies, antibody-drug conjugates, immunotoxins), vaccines, and CAR-T cell therapy.

The safety of CAR-T cells targeting MSLN in the treatment of cancers has also been verified in several clinical trials on lung cancers (NCT01583686, NCT02414269, NCT01355965). Professor Li Peng's group at the Chinese Academy of Science designed third generation CAR-T cells targeting MSLN and validated their use in both human PDAC cell lines, animal models, and in 4 patients with advanced malignancies. In a 42-year-old man with metastatic PDAC, the MSLN targeted CAR-T treatment led to complete response follow several hepatic artery infusion and intravenous infusion. These early cases confirmed the safety of these MSLN targeted CAR-T cells.

In the current proposed feasibility study, the researcher hypothesise that Endoscopic ultrasound (EUS)-guided injection of MSLN targeted CAR-T cells into PDAC can induce a tumor response, improve rate of R0 resection and translate into better patient survival.

DETAILED DESCRIPTION:
In the management of patients with PDAC, the role of neoadjuvant therapy is less certain. Neoadjuvant therapy for pancreatic cancer can in theory control early systemic spread and improve rate of R0 resection (2). In the ESPAC-5 study, neoadjuvant combination chemotherapy did not increase rate of resection who had borderline-resectable disease but appears to improve overall survival (OS) (3). The Charité Onkologie (CONKO-007) trial showed that the addition of radiation to chemotherapy improved R0 resection rate and complete pathological response (pCR) but did not impact on OS (4).

Chimeric antigen receptor (CAR) T-cell therapy may represent a new paradigm in the treatment of pancreatic cancer. Mesothelin (MSLN) is a 40 kDa membrane protein minimally expressed in normal cells, but highly expressed in a variety of cancer cells, such as mesothelioma, lung, breast, ovarian, gastric and pancreatic cancer. MSLN is expressed in about 80% of PDAC.

Mesothelin is the receptor of tumor antigen CA-125 (also known as MUC16). Tumor expressing CA-125 can combine with mesothelin on the surface of mesothelial cells in pleural or peritoneal cavity, resulting in increased cell adhesion and promoting metastatic diffusion (5). In pancreatic cancers, mesothelin plays a role in tumorigenesis by increasing cell proliferation, migration and S phase cell population. Its limited expression in normal human tissues and high expression in many cancers make it an attractive tumor-related antigen for cancer treatment (6).

There are several immunotherapies targeting MSLN for PDAC treatment, including antibody-based drugs (monoclonal antibodies, antibody-drug conjugates, immunotoxins), vaccines, and CART cell therapy. For example, the recombinant protein preparation SS1(dsFv)PE38 (SS1P), which is composed of high affinity Fv (variable fragment) targeting MSLN and Pseudomonas exotoxin A (PE) fusion, has entered clinical trials as a drug (7). There is also an antibody-drug conjugate, Anetumab ravtansine (BAY 94-9343), which is made by conjugating human anti-MSLN antibody with maytansinol tubulin inhibitor (DM4) through a connector containing disulfide bond. In vivo, anetumab ravtansine is specifically localized in tumors that express MSLN and inhibits the growth of pancreatic cancer, ovarian cancer, mesothelioma and other tumors. The safety of CAR-T cells targeting MSLN in the treatment of cancers has also been verified in several clinical trials on lung cancers (NCT01583686, NCT02414269, NCT01355965). Professor Li Peng's group at the Chinese Academy of Science designed third generation CAR-T cells targeting MSLN and validated their use in both human PDAC cell lines, animal models, and in 4 patients with advanced malignancies. In a 42-year-old man with metastatic PDAC, the MSLN targeted CAR-T treatment led to complete response following several hepatic artery infusion and intravenous infusion. These early cases confirmed the safety of these MSLN targeted CAR-T cells.

In the current proposed feasibility study, the researcher hypothesize that EUS-guided injection of MSLN targeted CAR-T cells into PDAC can induce a tumor response, improve rate of R0 resection and translate into better patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed pancreatic cancer planned for curative resection.
* Age 18 to 70 years old
* Measurable tumors according to RECIST 1.1s
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* A sufficient number of T cells taken through lymphopheresis (CD3+ T cells>1x109).
* Patients with preserved organ function as evidenced by
* Haematological: Hemoglobin ≥ 8g/dL; Platelet ≥ 75×109/L; INR≤1.5; Absolute neutrophil count (ANC) ≥ 1.5

  ×109 /L; Absolute lymphocyte count ≥ 0.4×109 /L
* Renal: Creatinine < 1.5 upper limit normal (ULN) mg/dL or Creatinine clearance ≥40 ml/min
* Bilirubin <1.5 ULN μmol/L; Alanine Aminotransferase (ALT) <3 IU/L; Albumin ≥30 g/L
* Willing and able to provide written, signed informed consent
* Sexually active subjects must be willing to use an acceptable method of contraception such as double barrier contraception during treatment and for 12 months after the last dose
* Females of childbearing potential must have a negative serum pregnancy test at screening and willing to have additional pregnancy tests during the study.
* Females considered non-childbearing potential include those who have been in menopause for at least 1 year or had tubal ligation at least 1 year prior to screening, or who have had total hysterectomy

Exclusion Criteria:

* Patients with AIDS
* Patients with serum HBsAg positive
* The patient has an active or uncontrolled infection.
* Subjects with severe heart, brain, liver, kidney or hematopoietic diseases, or psychosis who are not suitable for surgical resection
* In the first evaluation experiment, expansion ability of T cells activated by Cluster of Differentiation (CD) CD3/CD28 magnetic beads is less than 5 times.
* Pregnant or lactating women
* Those who participate in other clinical trials.
* History of chronic pancreatitis or Immunoglobulin G4 (IgG4) disease
* Patients who require splenectomy during surgery for pancreatic cancer. History of second malignancy except for any of the following:

( • Carcinoma in situ of the cervix or non-melanoma skin cancer ) ( • A cancer diagnosed and curatively treated ≥5 years prior to leukapheresis with no subsequent evidence of cancer recurrence )

* History of or waiting for organ transplantation, including liver transplantation
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
pathologic response | 3 months
  Proportion of major pathologic response on resected specimen of pancreatic tumour

SECONDARY OUTCOMES:
Radiological response | 4 weeks
  Radiological response according to RECIST 1.1 measured on CT 4 weeks after EUS guided MSLN CAR-T injection (i.e. tumor volumetric reduction at trial entry and 4 weeks after MSLN CAR-T injection).
Rate of R0 surgical resection | 3 months
  Rate of R0 surgical resection after EUS-guided injection of MSLN-targeted CAR-T cells
Serious Adverse Event | 1 year
  Incidence rate of serious adverse events of grade III and above.
Disease free and overall survival | 10 year
  Disease free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: James Lau, MD, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park W, Chawla A, O'Reilly EM. Pancreatic Cancer: A Review. JAMA. 2021 Sep 7;326(9):851-862. doi: 10.1001/jama.2021.13027. PMID 34547082
- [Background] Springfeld C, Ferrone CR, Katz MHG, Philip PA, Hong TS, Hackert T, Buchler MW, Neoptolemos J. Neoadjuvant therapy for pancreatic cancer. Nat Rev Clin Oncol. 2023 May;20(5):318-337. doi: 10.1038/s41571-023-00746-1. Epub 2023 Mar 17. PMID 36932224
- [Background] Ghaneh P, Palmer D, Cicconi S, Jackson R, Halloran CM, Rawcliffe C, Sripadam R, Mukherjee S, Soonawalla Z, Wadsley J, Al-Mukhtar A, Dickson E, Graham J, Jiao L, Wasan HS, Tait IS, Prachalias A, Ross P, Valle JW, O'Reilly DA, Al-Sarireh B, Gwynne S, Ahmed I, Connolly K, Yim KL, Cunningham D, Armstrong T, Archer C, Roberts K, Ma YT, Springfeld C, Tjaden C, Hackert T, Buchler MW, Neoptolemos JP; European Study Group for Pancreatic Cancer. Immediate surgery compared with short-course neoadjuvant gemcitabine plus capecitabine, FOLFIRINOX, or chemoradiotherapy in patients with borderline resectable pancreatic cancer (ESPAC5): a four-arm, multicentre, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):157-168. doi: 10.1016/S2468-1253(22)00348-X. Epub 2022 Dec 12. PMID 36521500
- [Background] Fietkau R, Ghadimi M, Grützmann R, Wittel UA, Jacobasch L, Uhl W, Croner RS, Bechstein WO, Neumann UP, Waldschmidt D, Boeck SH, Moosmann N, Reinacher-Schick AC, Golcher H, Adler W, Semrau S, Kallies A, Hecht M, Tannapfel A, Oettle H. Randomized phase III trial of induction chemotherapy followed by chemoradiotherapy or chemotherapy alone for nonresectable locally advanced pancreatic cancer: First results of the CONKO-007 trial. J Clin Oncol. 2022;40: issue 16 suppl.4008
- [Background] Chen SH, Hung WC, Wang P, Paul C, Konstantopoulos K. Mesothelin binding to CA125/MUC16 promotes pancreatic cancer cell motility and invasion via MMP-7 activation. Sci Rep. 2013;3:1870. doi: 10.1038/srep01870. PMID 23694968
- [Background] Kachala SS, Bograd AJ, Villena-Vargas J, Suzuki K, Servais EL, Kadota K, Chou J, Sima CS, Vertes E, Rusch VW, Travis WD, Sadelain M, Adusumilli PS. Mesothelin overexpression is a marker of tumor aggressiveness and is associated with reduced recurrence-free and overall survival in early-stage lung adenocarcinoma. Clin Cancer Res. 2014 Feb 15;20(4):1020-8. doi: 10.1158/1078-0432.CCR-13-1862. Epub 2013 Dec 13. PMID 24334761
- [Background] Hassan R, Bullock S, Premkumar A, Kreitman RJ, Kindler H, Willingham MC, Pastan I. Phase I study of SS1P, a recombinant anti-mesothelin immunotoxin given as a bolus I.V. infusion to patients with mesothelin-expressing mesothelioma, ovarian, and pancreatic cancers. Clin Cancer Res. 2007 Sep 1;13(17):5144-9. doi: 10.1158/1078-0432.CCR-07-0869. PMID 17785569
- [Background] Wang H, Chetty R, Hosseini M, Allende DS, Esposito I, Matsuda Y, Deshpande V, Shi J, Dhall D, Jang KT, Kim GE, Luchini C, Graham RP, Reid MD, Basturk O, Hruban RH, Krasinskas A, Klimstra DS, Adsay V; Pancreatobiliary Pathology Society. Pathologic Examination of Pancreatic Specimens Resected for Treated Pancreatic Ductal Adenocarcinoma: Recommendations From the Pancreatobiliary Pathology Society. Am J Surg Pathol. 2022 Jun 1;46(6):754-764. doi: 10.1097/PAS.0000000000001853. Epub 2021 Dec 15. PMID 34889852